CLINICAL TRIAL: NCT04566978
Title: A Pilot Study of 89Zr-DFO-REGN3767 Anti LAG-3 Antibody Positron Emission Tomography in Patients With Relapsed/Refractory DLBCL
Brief Title: 89Zr-DFO-REGN3767 in PET Scans in People With Diffuse Large B Cell Lymphoma (DLBCL)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-479
Record Dates: First submitted 2020-09-15; First posted 2020-09-28 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Large B-cell Lymphoma; DLBCL
Keywords: Large B-cell Lymphoma; DLBCL; Memorial Sloan Kettering Cancer Center; 19-479; 89Zr-DFO-REGN3767; anti LAG-3 antibody
MeSH Terms: interventions — Positron Emission Tomography Computed Tomography

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Up to 3 participants will be enrolled to receive a single dose of 89Zr-DFO-REGN3767 (total 2mg antibody mass). Participant to undergo 3 PET/CT scans and concurrent blood draws for PK
  Interventions: Drug: 89Zr-DFO-REGN3767; Diagnostic Test: PET/CT
- Cohort 2 (Experimental): Up to 3 participants will be enrolled to receive a total 5mg of 89Zr-DFO-REGN3767 (+REGN3767) total antibody mass for PK and serial imaging with 3 PET/CT scans
  Interventions: Drug: 89Zr-DFO-REGN3767; Diagnostic Test: PET/CT
- Cohort 3 (Experimental): Up to 3 participants will be enrolled to receive a total 10mg of 89Zr-DFO-REGN3767 (+REGN3767) total antibody mass for PK and serial imaging with 3 PET/CT scans
  Interventions: Drug: 89Zr-DFO-REGN3767; Diagnostic Test: PET/CT
- Cohort 4 (Experimental): Up to 3 participants will be enrolled to receive a total 20mg of 89Zr-DFO-REGN3767 (+REGN3767) total antibody mass for PK and serial imaging with 3 PET/CT scans
  Interventions: Drug: 89Zr-DFO-REGN3767; Diagnostic Test: PET/CT

INTERVENTIONS:
Drug: 89Zr-DFO-REGN3767 — 89Zr-DFO-REGN3767 is comprised of the anti-LAG-3 antibody, REGN3767 labeled with the positron-emitter zirconium-89 (89Zr) through the chelator-linker DFO. REGN3767 is an investigational monoclonal antibody that target LAG-3 receptors.
Diagnostic Test: PET/CT — A PET/CT scan extending from top of skull to feet will be performed to determine the biodistribution.
  Part A patients will be imaged at three time points post-injection to allow for selection of optimal imaging time and dosimetry determination. For these patients, top of skull to feet scans will be acquired:
  * Within one to four hours following injection of tracer on Day 1
  * 24-72 hours post-injection (Day 2-4)
  * 20-168 hours post-injection (once during days 5-7)

SUMMARY:
The main purposes of this study include:

Looking at the way the body absorbs, distributes, and gets rid of 89Zr-DFO-REGN3767

Finding the best dose amount of 89Zr-DFO-REGN3767

Finding the best time for PET scanning after injection of 89Zr-DFO-REGN3767

ELIGIBILITY:
Inclusion Criteria:

A patient must be eligible for DLBCL expansion cohort 9 in study 17-421 and, in addition, meet the following criteria to be eligible for inclusion in the study:

* Measurable disease by Lugano criteria, with at least one lesion outside of the liver
* Patients must have eGFR >50 mL/min/1.73m2.

Exclusion Criteria:

A patient must be eligible for DLBCL expansion cohort 9 in study 17-421 and, in addition, a patient who meets any of the following criteria will be excluded from the study:

* Patients who have permanently discontinued anti-cancer immune modulating therapies due to drug-related toxicity.
* Has not yet recovered (i.e. ≤ Grade 1 or baseline) from any acute toxicities from prior anticancer therapy except for laboratory changes as described in inclusion criteria in study 17-421, except as noted. NOTE: Patients with chronic or stable toxicity following approved therapy, such as mild persistent neuropathy, are allowed.
* Has received radiation therapy within 14 days of first administration of study drug or has not recovered (i.e. ≤ Grade 1 or baseline) from adverse events, except for laboratory changes as described in inclusion criteria, except as noted. NOTE: Patients with chronic or stable toxicity, such as mild persistent neuropathy, are allowed.
* Women who are pregnant, breastfeeding *Postmenopausal women must be amenorrhoeic for at least 12 months in order not to be considered of childbearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation. Pregnancy testing and screening will be performed per MSK and Department of Radiology standard pregnancy screening guidelines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-09-11 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

PRIMARY OUTCOMES:
Biodistribution of 89Zr-DFO-REGN3767 | 2 years
  A PET/CT scan extending from top of skull to feet will be performed to determine the biodistribution of 89Zr-DFO-REGN3767
Optimal 89Zr-DFO-REGN3767 mass dose for tumor targeting | 2 years
  Determine the optimal 89Zr-DFO-REGN3767 mass dose for tumor targeting
Optimal time for imaging and tumor uptake post 89Zr-DFO-REGN3767 administration | 2 years
  Determine the optimal time for imaging and tumor uptake post 89Zr-DFO-REGN3767 administration
Tumor lesion uptake of 89Zr-DFO-REGN3767 and correlate with LAG-3 expression by IHC | 2 years
  Evaluate tumor lesion uptake of 89Zr-DFO-REGN3767 and correlate with LAG-3 expression by IHC in tumors will be compared descriptively with other biomarkers of tumor immune environment characterized in biopsies, such as quantitation of IHC score (LAG-3 and / or other immune cell markers), or other biomarker measures.

CONTACTS AND LOCATIONS:
Overall Officials: Neeta Pandi-Taskar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org